CLINICAL TRIAL: NCT01094509
Title: Tai Chi and Guided Autobiography for Remediation of Age-related Cognitive Decline
Brief Title: Activities for Cognitive Enhancement of Seniors
Acronym: ACE-Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Victor W. Henderson, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SU-02042010-4903; R01AG034639 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Aging
MeSH Terms: interventions — Tai Ji; Qigong

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Tai Chi (Experimental): Tai Chi exercises
  Interventions: Behavioral: Tai Chi
- Guided autobiography (Experimental): Autobiographical writing during class sessions and at home
  Interventions: Behavioral: Guided autobiography
- Qigong (Experimental): Qigong exercises (exploratory, not part of the original protocol, added to gain experience with this intervention)
  Interventions: Behavioral: Qigong
- Successful aging (Active Comparator): Seminars on the theme of successful aging
  Interventions: Behavioral: Successful aging
- Combination (Experimental): Combination of Tai Chi exercises and autobiographical writing
  Interventions: Behavioral: Combination
- Comparison (Placebo Comparator): No assigned experimental activity (exploratory, not part of the original protocol, added to gain experience with a placebo comparator)
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi classes and exercises
  Arms: Tai Chi
Behavioral: Guided autobiography — Autobiographical writing in class and at home
  Arms: Guided autobiography
Behavioral: Qigong — Qigong classes and exercises (exploratory)
  Arms: Qigong
Behavioral: Successful aging — Seminar series on the theme of successful aging
  Arms: Successful aging
Behavioral: Combination — Combination of Tai Chi exercises and autobiographical writing
  Arms: Combination
Behavioral: Comparison — No assigned behavioral activity (exploratory)
  Arms: Comparison

SUMMARY:
Cognitive aging and cognitive decline are important public health concerns in an aging US population. The investigators will conduct a randomized controlled trail among healthy older adults to assess effects of several innovative activities on remediation of age-related cognitive decline.

DETAILED DESCRIPTION:
ACE-Seniors is designed as a single-site trial of four randomly assigned interventions, Tai Chi exercise, autobiographical writing, both Tai Chi and autobiography (dual intervention), and general health education. Participants are relatively healthy adults aged 70 years or older, who are not regular practitioners of Tai Chi or regular writers. They are without medical or neurological disorders that would substantially limit the ability to participate in study interventions, without dementia or mild cognitive impairment, relatively sedentary, able to walk unassisted, and able to score 4 or better on the Short Physical Performance Battery. Interventions are administered over a 6 month period of time, with similar exposure times among the four groups. The prespecified primary endpoint is derived from a composite neuropsychological measure, based on three tests of executive function and three tests of episodic memory. The planned sample size is 96 (24 per group). Intention-to-treat analysis will include all eligible participants who complete baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older.
* No other household member already enrolled.
* In reasonably good health: no serious cognitive problem; free of any condition that would limit your ability to participate in Tai Chi classes (a moderate intensity exercise), in Qigong exercises, in a writing program, or in a seminar series.
* Not presently engaged in a regular exercise program; not presently engaged in Tai Chi Qigong or another form of Eastern exercise; and not a regular writer.
* Not now engaged in research to enhance cognitive skills.
* Willing to travel to Stanford for ACE-Seniors program classes. Planning to be in the area during most of the coming year;
* Willing to be assigned randomly (by chance) to one of the ACE-Senior activities.

Exclusion Criteria:

* Failure to meet inclusion criteria.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 175 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cognitive (executive function and episodic memory) | 6 and 12 months

SECONDARY OUTCOMES:
Other cognitive measures | 6 and 12 months
Physical performance and other non-cognitive measures | 6 and 12 months
Adherence and retention | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Victor Henderson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States